CLINICAL TRIAL: NCT01118663
Title: A Multi-center, Double-blind, Randomized, Controlled Study to Determine the Efficacy and Safety of a New Formulation of Acetylcysteine Injection
Brief Title: Safety and Efficacy Study of a New Formulation of Acetylcysteine Injection
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Cumberland Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CPI-NAC-001
Record Dates: First submitted 2010-05-04; First posted 2010-05-07 (Estimated); Results first posted 2014-08-04 (Estimated); Last update posted 2014-08-04 (Estimated); Status verified 2014-08

CONDITIONS: Acetaminophen Overdose
Keywords: Acetaminophen overdose; induced hepatotoxicity, liver injury
MeSH Terms: interventions — Edetic Acid; Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Acetadote without EDTA (Experimental): Acetadote EF [Ethylenediaminetetraacetic Acid (EDTA) - Free]
  Interventions: Drug: Acetadote EF (Ethylenediaminetetraacetic Acid (EDTA) - Free)
- Acetadote (Active Comparator): Acetadote [Old formulation containing EDTA]
  Interventions: Drug: Acetadote

INTERVENTIONS:
Drug: Acetadote EF (Ethylenediaminetetraacetic Acid (EDTA) - Free) — Acetadote EF (Ethylenediaminetetraacetic Acid (EDTA) - Free) {new formulation} 200 mg/kg in 1000 ml diluent over 4 hours; then 100 mg/kg in 1000 ml diluent over 16 hours
  Other Names: acetylcysteine
  Arms: Acetadote without EDTA
Drug: Acetadote — Acetadote [old formulation] 150 mg/kg in 200 mL diluent over 60 minutes; then Acetadote 50 mg/kg in 500 mL diluent over 4 hours; then Acetadote 100 mg/kg in 1000 mL diluent over 16 hours.
  Other Names: acetylcysteine
  Arms: Acetadote

SUMMARY:
The primary purpose of this study is determine if a new formulation of Acetadote is at least as effective as the current formulation in the prevention and treatment of acetaminophen overdose related liver injury.

DETAILED DESCRIPTION:
The primary objective of this study is to demonstrate non-inferiority of efficacy determined by the proportion of subjects who develop hepatotoxicity when treated with a new formulation of Acetadote and the proposed new dosing regimen compared to the rate of hepatotoxicity with the current formulation of Acetadote and the current dosing regimen.

ELIGIBILITY:
Inclusion Criteria:

1) Any subject requiring treatment with acetylcysteine for acute acetaminophen toxicity

Exclusion Criteria:

1. History of allergy or hypersensitivity to acetylcysteine or any component of Acetadote.
2. Exposed to investigational drugs within 30 days before Clinical Trial Material (CTM) administration.
3. Pregnant or nursing.
4. Less than 12 years of age.
5. Have a baseline alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >1000 U/L.
6. Have a baseline International Normalized. Ratio (INR) > 2.0
7. Be on dialysis or having existing renal injury such that the volume of the study drug administration would render the patient unsuitable for the study, in the opinion of the investigator.
8. Have congestive heart failure such that the volume of the study drug administration would render the patient unsuitable for the study, in the opinion of the investigator.
9. Inability to understand the requirements of the study. Subjects must be willing to provide written informed consent or consent of parent/legal guardian (as evidenced by signature on an informed consent document approved by an Institutional Review Board [IRB]), and agree to abide by the study restrictions. (If the subject is incapacitated, informed consent will be sought from a legally acceptable representative).
10. Refusal to provide written authorization for use and disclosure of protected health information.
11. Be otherwise unsuitable for the study, in the opinion of the Investigator.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2010-09; Primary Completion 2012-11 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Art Wheeler, MD, Study Director — Cumberland Pharmaceuticals, Inc.
Locations (14):
- United States (14):
  - Maricopa Medical Center, Phoenix, Arizona
  - Loma Linda University Medical Center, Loma Linda, California
  - University of California Irvine Medical Center, Orange, California
  - UCSD Medical Center, San Diego, California
  - University of Colorado Hospital, Aurora, Colorado
  - Denver Health and Hospital Authority, Denver, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - LSU Health Sciences Center - Shreveport, Shreveport, Louisiana
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - UMass Memorial Medical Center, Worcester, Massachusetts
  - Spectrum Health Butterworth Hospital, Grand Rapids, Michigan
  - East Carolina University Medical Center, Greenville, North Carolina
  - Toledo Hospital, Toledo, Ohio
  - Scott & White Medical Center, Temple, Texas

REFERENCES:
- [Background] Bhushan M, Beck MH. Allergic contact dermatitis from disodium ethylenediamine tetra-acetic acid (EDTA) in a local anaesthetic. Contact Dermatitis. 1998 Mar;38(3):183. doi: 10.1111/j.1600-0536.1998.tb05702.x. No abstract available. PMID 9536427
- [Background] van Laar T, van Hilten B, Neef C, Rutgers AW, Pavel S, Bruijn JA. The role of EDTA in provoking allergic reactions to subcutaneous infusion of apomorphine in patients with Parkinson's disease: a histologic study. Mov Disord. 1998 Jan;13(1):52-5. doi: 10.1002/mds.870130113. PMID 9452326
- [Background] Kimura M, Kawada A. Contact dermatitis due to trisodium ethylenediaminetetra-acetic acid (EDTA) in a cosmetic lotion. Contact Dermatitis. 1999 Dec;41(6):341. doi: 10.1111/j.1600-0536.1999.tb06184.x. No abstract available. PMID 10617216
- [Background] Marik PE. Propofol: therapeutic indications and side-effects. Curr Pharm Des. 2004;10(29):3639-49. doi: 10.2174/1381612043382846. PMID 15579060

RESULTS

PARTICIPANT FLOW:
Groups:
- Acetadote Without EDTA: Acetadote EF [Ethylenediaminetetraacetic Acid (EDTA) - Free]
  Acetadote EF [Ethylenediaminetetraacetic Acid (EDTA) - Free]: Acetadote EF [Ethylenediaminetetraacetic Acid (EDTA) - Free] {new formulation} 200 mg/kg in 1000 ml diluent over 4 hours; then 100 mg/kg in 1000 ml diluent over 16 hours
Period: Overall Study
Arm/Group | Acetadote Without EDTA | Acetadote
Started | 7 | 10
Completed | 5 | 8
Not Completed | 2 | 2
Not completed — Adverse Event | 2 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Acetadote Without EDTA | Acetadote | Total
Number analyzed (Participants) | 7 | 10 | 17
Age, Customized [Number; unit: participants]
  ≤ 18 years | 1 | 0 | 1
  19-59 years | 6 | 8 | 14
  ≥ 60 years | 0 | 2 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 7 | 12
  Male | 2 | 3 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 6
  Not Hispanic or Latino | 4 | 7 | 11
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 6 | 9 | 15
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 7 | 10 | 17

OUTCOME MEASURES:

1. Primary Outcome: The Incidence of Hepatoxicity as Measured by the Percentage of Subjects With an Alanine Transaminase (ALT) or Aspartate Transaminase (AST) Value > 1000 U/L Versus Those With an ALT and AST < 1000 U/L
Description: Because the study was terminated prematurely due to lack of enrollment, there was an insufficient sample size to conduct an efficacy analysis.
Time Frame: 21 hours
Population: Because the study was terminated prematurely due to lack of enrollment, there was insufficient sample size to conduct efficacy analysis.
Arm/Group | Acetadote Without EDTA | Acetadote
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: To Evaluate the Percentage of Subjects Requiring Continued Therapy
Description: as for outcome 1
Time Frame: 21 hours
Population: as for outcome 1
Arm/Group | Acetadote Without EDTA | Acetadote
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: To Evaluate the Incidence of Clinical Need for Therapy Beyond the Current 21 Hour FDA Approved Dosing Regimen.
Description: as for outcome 1
Time Frame: 42 hours
Population: as for outcome 1
Arm/Group | Acetadote Without EDTA | Acetadote
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: To Evaluate the Incidence of Treatment Emergent Adverse Events
Time Frame: 21-42 hours
Measure: Number; unit: Number of Events
Arm/Group | Acetadote Without EDTA | Acetadote
Number analyzed (Participants) | 7 | 10
Number of Events | 13 | 14

5. Secondary Outcome: To Evaluate the Incidence of Anaphylactoid Reaction.
Description: Data analysis was conducted on the subjects enrolled in the study prior to study termination. Because the study was terminated prematurely due to lack of enrollment, there was an insufficient sample size to conduct an efficacy analysis.
Time Frame: 1 hour
Measure: Number; unit: participants
Arm/Group | Acetadote Without EDTA | Acetadote
Number analyzed (Participants) | 7 | 10
participants | 0 | 1

ADVERSE EVENTS:
Arm/Group | Acetadote Without EDTA | Acetadote
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/10
Other Adverse Events (participants affected / at risk) | 5/7 | 7/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Acetadote Without EDTA (N=7) | Acetadote (N=10)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Flushing (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Blood Potassium Decreased (Investigations) | 0 (0) | 1 (1)
Livedo Reticularis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (2)
Vomiting (Gastrointestinal disorders) | 3 (3) | 3 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chest Discomfort (General disorders) | 0 (0) | 1 (1)
Anaphylactoid Reaction (Immune system disorders) | 0 (0) | 1 (1)
Chest Pain (General disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Blood Magnesium Decreased (Investigations) | 1 (1) | 0 (0)
Trismus (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Abdominal Discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No